CLINICAL TRIAL: NCT01437605
Title: A Randomized Phase II Study to Assess the Safety and Immunogenicity of recMAGE-A3+AS15 ASCI With or Without Poly IC:LC in Patients With Resected MAGE-A3 Positive, Stage IV Melanoma
Brief Title: Phase II Study to Assess the Safety and Immunogenicity of recMAGE-A3+AS15 ASCI With or Without Poly IC:LC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Treatment Ineffective
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: GlaxoSmithKline (Industry); Oncovir, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16545
Record Dates: First submitted 2011-09-19; First posted 2011-09-21 (Estimated); Results first posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Melanoma
Keywords: Resected; Skin; Stage IV
MeSH Terms: conditions — Melanoma | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: recMAGE-A3 + AS15 (Active Comparator): ASCI injections without Poly IC:LC
  Interventions: Drug: MAGE-A3 ASCI injections without Poly IC:LC
- B: recMAGE-A3 + AS15 + Poly IC:LC (Active Comparator): ASCI injections with Poly IC:LC
  Interventions: Drug: MAGE-A3 ASCI injections with Poly IC:LC

INTERVENTIONS:
Drug: MAGE-A3 ASCI injections without Poly IC:LC — MAGE-A3 ASCI injections without Poly IC:LC as outlined in Detailed Description
  Other Names: Recombinant MAGE-A3 protein; AS15 adjuvant
  Arms: A: recMAGE-A3 + AS15
Drug: MAGE-A3 ASCI injections with Poly IC:LC — MAGE-A3 ASCI injections with Poly IC:LC as outlined in Detailed Description
  Other Names: Recombinant MAGE-A3 protein; AS15 adjuvant; Hiltonol; NSC 301463
  Arms: B: recMAGE-A3 + AS15 + Poly IC:LC

SUMMARY:
The overall purpose of this research study is to find a better way to treat melanoma.

The goals of this study are:

1. To measure the side effects of and find out how well patients tolerate the recMAGE-A3 + AS15 ASCI (MAGE-A3 ASCI) treatment with or without the Poly IC:LC
2. To see how well the patient's immune system responds to the MAGE-A3 ASCI treatment with or without the Poly IC:LC
3. To measure the rate of return of the patient's tumor after the MAGE-A3 ASCI treatment with or without the Poly IC:LC
4. To measure the rate of return of the patient's tumor in two groups of patients: one group positive for the gene signature, and the other group not positive for the gene signature in their tumor after the MAGE-A3 ASCI treatment with or without the Poly IC:LC.

DETAILED DESCRIPTION:
In the first year, participants may receive up to 8 injections given in the following order:

1. 5 ASCI injections with or without Poly IC:LC with a 3-week interval between each.
2. 3 ASCI injections with or without Poly IC:LC with a 3-month interval between each.

   During years 2 through 3, participants may receive up to 5 ASCI injections with or without Poly IC:LC given in the following order:
3. During year 2, ASCI injections with or without Poly IC:LC will be given every 3 months for a total of up to 3 injections.
4. During year 3, ASCI injections with or without Poly IC:LC will continue to be given every 3 months for a total of up to 2 more injections.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for the study will be obtained prior to the performance of MAGE-A3 expression screening on resected tumor tissue or any other protocol-specific procedure.
* Male or female patient with histologically proven and completely resected stage IV cutaneous or mucosal melanoma. In terms of the American Joint Committee on Cancer (AJCC) classification [AJCC, 2009], this means that patients with resected M1a-b-c (stage IV) disease may be enrolled.
* The patient must have been surgically rendered free of disease no more than 12 weeks before the randomization.
* Patient is equal to or greater than 18 years old at the time of signing the informed consent form.
* The patient's tumor shows expression of the MAGE-A3 gene, as determined by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) analysis on paraffin imbedded tumor tissue (FFPE). In all patients in whom it can be obtained, a frozen portion of the resected tumor will be analyzed for gene profiling.
* The patient has fully recovered from surgery.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at the time of randomization.
* The patient must have adequate bone-marrow reserve, adequate renal function and adequate hepatic function as assessed by standard laboratory criteria: Absolute neutrophil count (ANC) equal to or greater than 1.5 x 10^9/L, Platelet count equal to or greater than 75 x 10^9/L, Serum creatinine equal to or less than 1.5 times the Upper Limit of Normal (ULN), Total bilirubin equal to or less than 1.5 times the ULN, Transaminase (ALT - AST) equal to or less than 2.5 times the ULN
* If the patient is female, she must be of non-childbearing potential, i.e. have a current tubal ligation, hysterectomy, ovariectomy or be post menopausal, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to randomization, have a negative pregnancy test and continue such precautions during the entire study treatment period and for 2 months after completion of the injection series.
* Men must also agree to use an adequate method of contraception.
* In the opinion of the investigator, the patient can and will comply with all the requirements of the protocol.

Exclusion Criteria:

* The patient has an ocular melanoma.
* The patient has in-transit metastases.
* The patient has been treated or is scheduled to be treated with an adjuvant anticancer therapy after the metastasectomy that qualifies the patient for inclusion in the present trial.
* One prior systemic treatment with an immunomodulator (i.e., interferon, vaccine and/or anti-CTLA-4) after a previous surgery is permitted, provided that the last dose has been administered at least 45 days before randomization in the present trial.
* Previous radiotherapy is permitted, provided that the treatment has been completed before the surgery that qualifies the patient for participation in the present trial.
* The patient requires concomitant chronic treatment (more than 7 consecutive days) with systemic corticosteroids or any other immunosuppressive agents. The use of prednisone, or equivalent, at a dose of < 0.125 mg/kg/day (absolute maximum 10 mg/day) or topical steroids is permitted.
* Use of any investigational or non-registered product (drug or vaccine) other than the study treatment within 30 days preceding the randomization or planned use during the study period.
* The patient has a history of autoimmune disease such as, but not limited to, multiple sclerosis, lupus, and inflammatory bowel disease. Patients with vitiligo are not excluded.
* The patient has a family history of congenital or hereditary immunodeficiency.
* The patient is known to be positive for Human Immunodeficiency Virus (HIV) or has another confirmed or suspected immunosuppressive or immunodeficient condition.
* History of allergic disease or reactions likely to be exacerbated by any component of the treatments.
* The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent or to comply with the trial procedures.
* The patient has concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
* The patient has previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers or carcinoma in situ of the cervix or effectively treated malignancy that has been in remission for over 5 years and is highly likely to have been cured.
* The patient has an uncontrolled bleeding disorder.
* For female patients: the patient is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-10-11 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Khushalani, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A: recMAGE-A3 + AS15 | B: recMAGE-A3 + AS15 + Poly IC:LC
Started | 9 | 5
Completed | 9 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants enrolled on study. All participants who received study treatment. Outcome Measures: All participants evaluable at time of analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | A: recMAGE-A3 + AS15 | B: recMAGE-A3 + AS15 + Poly IC:LC | Total
Number analyzed (Participants) | 9 | 5 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 3 | 11
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 7 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race White / Ethnicity Non-Hispanic | 9 | 5 | 14
Region of Enrollment [Number; unit: participants]
  United States | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Related to Study Treatment
Description: Number of participants with adverse events after receiving one dose of recMAGE-A3 + AS15 ASCI or recMAGEA3 + AS15 ASCI in combination with Poly IC:LC
Time Frame: Beginning of Treatment to End of Follow Up - up to 5 years per participant
Measure: Count of Participants; unit: Participants
Arm/Group | A: recMAGE-A3 + AS15 | B: recMAGE-A3 + AS15 + Poly IC:LC
Number analyzed (Participants) | 9 | 5
Participants | 9 | 5

2. Secondary Outcome: Immunogenicity Per Treatment Arm
Description: Laboratory Endpoint: Assessment of the immunogenicity of the two regimens. Serum antibodies (such as Anti-MAGE-A3) seropositivity status (a seropositive patient is a patient whose titre is greater than or equal to the cut-off value) will be the primary immune endpoints assessed. Seropositivity will be assessed at baseline, after 2, 4, 6, 7 and 9 administrations, post-treatment (i.e., at concluding visit) and one year after concluding visit (i.e., at follow-up visit 2).
Time Frame: Beginning of Treatment to End of Follow Up - up to 5 years per participant
Population: Data not collected (likely futility from low numbers enrolled when the protocol was closed to accrual)
Arm/Group | A: recMAGE-A3 + AS15 | B: recMAGE-A3 + AS15 + Poly IC:LC
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants With Relapse-Free Survival (RFS)
Description: RFS, defined as the time from randomization to the date of first relapse of melanoma or of death, whichever comes first. Percentage of participants with RFS, assessed up to 2 years is reported
Time Frame: Beginning of Treatment to End of Follow Up - up to 2 years per participant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A: recMAGE-A3 + AS15 | B: recMAGE-A3 + AS15 + Poly IC:LC
Number analyzed (Participants) | 9 | 5
percentage of participants
  1 Year RFS | 56 [20 to 80] | 40 [5 to 75]
  2 Year RFS | 33 [8 to 62] | 40 [5 to 75]

4. Secondary Outcome: Median Overall Survival (OS)
Description: OS defined as the interval from randomization to the date of death, irrespective of the cause of death; patients still alive will be censored at the date of the last assessment. The primary analysis will be based on the adjusted Cox regression model.
Time Frame: At 5 years
Population: Data not collected (likely futility from low numbers enrolled when the protocol was closed to accrual)
Arm/Group | A: recMAGE-A3 + AS15 | B: recMAGE-A3 + AS15 + Poly IC:LC
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Immunogenicity as Measured by T Cell Responses
Description: Immunogenicity as measured by T cell responses directed against MAGE-A3 antigen.
Time Frame: Beginning of Treatment to End of Follow Up - up to 5 years per participant
Population: Participants not analyzed due to low number of patients accrued to this study before closure for likely futility from other negative trials of MAGE-A3
Arm/Group | A: recMAGE-A3 + AS15 | B: recMAGE-A3 + AS15 + Poly IC:LC
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Correlation Between Gene Expression Profile and Treatment Clinical Activity
Description: A potential correlation between gene expression profile and treatment clinical activity (RFS) in both study arms (recMAGE-A3 + AS15 ASCI and recMAGE-A3 + AS15 ASCI in combination with Poly IC:LC).
Time Frame: Beginning of Treatment to End of Follow Up - up to 5 years per participant
Population: as for outcome 5
Arm/Group | A: recMAGE-A3 + AS15 | B: recMAGE-A3 + AS15 + Poly IC:LC
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 years and 11 months
Arm/Group | A: recMAGE-A3 + AS15 | B: recMAGE-A3 + AS15 + Poly IC:LC
All-Cause Mortality (participants affected / at risk) | 4/9 | 2/5
Serious Adverse Events (participants affected / at risk) | 3/9 | 1/5
Other Adverse Events (participants affected / at risk) | 9/9 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: recMAGE-A3 + AS15 (N=9) | B: recMAGE-A3 + AS15 + Poly IC:LC (N=5)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Infections and Infestations - Other, Specify (Infections and infestations) | 1 (1) | 0 (0)
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thromboembolic Event (Vascular disorders) | 1 (1) | 0 (0)
Central Nervous System Necrosis (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: recMAGE-A3 + AS15 (N=9) | B: recMAGE-A3 + AS15 + Poly IC:LC (N=5)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0)
Endocrine Disorders - Other, Specify (Endocrine disorders) | 0 (0) | 1 (2)
Blurred Vision (Eye disorders) | 1 (1) | 1 (1)
Dry Eye (Eye disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal Disorders - Other, Specify (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 2 (2) | 0 (0)
Edema Limbs (General disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 6 (17) | 3 (6)
Fever (General disorders) | 7 (14) | 3 (10)
Flu Like Symptoms (General disorders) | 5 (9) | 3 (3)
General Disorders and Administration Site Conditions - Other, Specify (General disorders) | 3 (5) | 0 (0)
Injection Site Reaction (General disorders) | 7 (20) | 4 (13)
Malaise (General disorders) | 1 (4) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Infections and Infestations - Other, Specify (Infections and infestations) | 0 (0) | 1 (1)
Papulopustular Rash (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Skin Infection (Infections and infestations) | 1 (2) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (2) | 0 (0)
Platelet Count Decreased (Investigations) | 1 (1) | 0 (0)
Weight Gain (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms Benign, Malignant and Unspecified (includes Cysts and Polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1)
Central Nervous System Necrosis (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 2 (3)
Headache (Nervous system disorders) | 6 (10) | 0 (0)
Memory Impairment (Nervous system disorders) | 1 (1) | 0 (0)
Nervous System Disorders - Other, Specify (Nervous system disorders) | 1 (3) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral Motor Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Spasticity (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Renal and Urinary Disorders - Other, Specify (Renal and urinary disorders) | 0 (0) | 1 (2)
Irregular Menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory, Thoracic and Mediastinal Disorders - Other, Specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail Loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Scalp Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and Subcutaneous Tissue Disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (2)
Hot Flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (3) | 0 (0)
Thromboembolic Event (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT01437605/Prot_SAP_000.pdf